CLINICAL TRIAL: NCT04300335
Title: The Feasibility and Effects of an Individualized Aerobic and Resistance Training Protocol for Patients Suffering From Multiple Myeloma With Varying Risk of Fall and Fracture - a Pilot Study
Brief Title: The Feasibility and Effects of Exercise on Patients Suffering From Multiple Myeloma
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was not started because the necessary resources could not yet be secured after COVID-19, which was the reason for the initial interruption of the study.
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Richard Crevenna, Univ.-Prof. Dr. Richard Crevenna, MBA, MMSc, Head of the Department of Physical Medicine, Rehabilitation and Occupational Medicine, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2172/2019
Record Dates: First submitted 2020-03-02; First posted 2020-03-09 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma
Keywords: exercise; fracture risk
MeSH Terms: conditions — Multiple Myeloma; Motor Activity

STUDY DESIGN:
Intervention Model Description: Group 1: Individual exercise prescription (high fracture risk and/or high risk of fall patients) Group 2: Group exercise (low fracture risk and low risk of fall patients)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Risk - Individual Exercise (Experimental): Patients who show an increased fracture risk and/or increased risk of fall in the screening assessments and are therefore allocated to an individualized personal training.
  Interventions: Other: Individual Exercise
- Low Risk - Group Exercise (Experimental): Patients who show neither increased fracture risk nor increased risk of fall in the screening assessments and are therefore allocated to the exercise group.
  Interventions: Other: Group Exercise

INTERVENTIONS:
Other: Individual Exercise — Supervised body weight & resistance band resistance exercises in a one-on-one personal training setting plus home based aerobic exercise
  Arms: High Risk - Individual Exercise
Other: Group Exercise — Supervised body weight & resistance band resistance exercises in a Group setting plus home based aerobic exercise
  Arms: Low Risk - Group Exercise

SUMMARY:
Multiple myeloma is the second most common haematological cancer with a cancer incidence of around 500 new cases in Austria per year . Novel treatment methods have significantly increased the cancer-specific survival rate in patients with multiple myeloma. For Austria, this means that 5- and 10-year survival rates rose from 32.1 to 46.4% and from 19.0 to 25.6% from the end of the 1980s to the end of the 2000s.

Longer survival is associated with the need to maintain independence and quality of life in the longer term. In this context, regular physical training has seen a significant increase in the importance of cancer in recent years.The guidelines of the American College of Sports Medicine still contain very general training recommendations for cancer patients. Either 150 minutes of moderate or 75 minutes of intensive endurance training per week are recommended, supplemented by at least two units of strengthening training and stretching exercises for the large muscle groups.

In a recent cross-sectional and pilot study with multiple myeloma patients that was carried out at the Clinic for Physical Medicine, Rehabilitation and Occupational Medicine at the Medical University of Vienna (EK 1725/2018), it was on the one hand identified that there was a discrepancy between these patients on the one hand has given actual and perceived risk of falling, and on the other hand it is concluded that training recommendations should be carried out separately in group and individual training according to the actual risk of falling and fracture.

The present project is the follow-up to this cross-sectional investigation. The aim is to examine the feasibility and effects of a structured, physical training program carried out over a period of 12 weeks on physical performance, quality of life, body composition and the risk of falling. The effects of patients with increased risk in individual training sessions are compared to those of lower risk patients in group training sessions. Furthermore, the study patients will be able to bring training partners with them to their own training units if available and for their own security. They are evaluated separately according to qualitative criteria.

DETAILED DESCRIPTION:
The aim of this study is to investigate the feasibility and effectiveness of individualized training support for multiple myeloma patient populations divided into high and low risk according to their fall and fracture risk. The primary hypothesis is that multiple myeloma patients who meet the criteria for a high risk of falling and / or fracture can achieve equivalent adherence rates and training effects through individually compiled individual training, such as multiple myeloma patients with low risk of falling who conduct group training.

The adherence rates are recorded via attendance lists for training and video conferences as well as a training diary for independent training. To record the training effects, physical performance and functionality are measured and the quality of life, sexuality, depression, fatigue, sleep quality, work ability and risk of falling are assessed using standardized, validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Myeloma after primary Treatment
* Sufficient knowledge of the German language to being able to follow the study procedures
* Cardiologic-internal clearance for exercise

Exclusion Criteria:

* Fulfillment of absolute exclusion criteria of the cardiovascular system or on the musculoskeletal system with regard to physical trainability
* Insufficient language knowledge
* Cognitively unable to follow the course of the study
* Severe mental illness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility (Adherence) | Adherence rates through 12 weeks of exercise intervention program
  We hypothesize that the adherence of "High Risk Patients" to a personal, individualized exercise intervention is equal to that of "Low Risk Patients" performing group exercise.

SECONDARY OUTCOMES:
VO2max | Baseline + 12 weeks
  Maximum oxygen consumption in a cardiopulmonary exercise testing
Handgrip Strength (HGS) | Baseline + 12 weeks
  Handgrip Dynamometer (JAMAR)
Six Minute Walk Test (6MWT) | Baseline + 12 weeks
  Distance covered when walking as fast as possible in six minutes
Tinetti-Test/Performance Oriented Mobility Assessment (POMA) | Baseline + 12 weeks
  Risk of Fall Assessment
Timed up and Go Test (TUG) | Baseline + 12 weeks
  Risk of Fall Assessment
Bioimpedance Analysis (BiA) | Baseline + 12 weeks
  Body Composition measurement measured with Nutribox (BiA)
Five Repetitions Sit-to-Stand Test (5STS) | Baseline + 12 weeks
  Test for Lower Extremity Strength (time needed to stand up and sit down on a chair 5 times)

OTHER OUTCOMES:
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Basic Module (EORTC QLQ-C30) | Baseline + 12 weeks
  Cancer specific quality of life (Questionnaire); Score range from 0 to 100; A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Myeloma Module (EORTC QLQ-MY20) | Baseline + 12 weeks
  Multiple myeloma specific quality of life (Questionnaire); Score range from 0 to 100; A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Fatigue Module (EORTC QLQ-FA12) | Baseline + 12 weeks
  Cancer related fatigue specific quality of life (Questionnaire); Score range from 0 to 100; A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Sexual Health Quality Module (EORTC QLQ-SHQ22) | Baseline + 12 weeks
  Cancer related sexual health specific quality of life (Questionnaire); Score range from 0 to 100; A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
International Physical Activity Questionnaire (IPAQ) | Baseline + 12 weeks
  Physical Activity (Questionnaire); Patients are asked about the frequency and volume of at least 10 minutes long episodes of vigorous and moderate physical activity during their last 7 days.
  Higher values indicate higher levels of physical activity.
Hospital Anxiety and Depression Scale (HADS) | Baseline + 12 weeks
  Anxiety and Depression (Questionnaire); Score range from 0-21; lower scores indicating lower levels anxiety and depression
Work Ability Index (WAI) | Baseline + 12 weeks
  Work Ability (Questionnaire); Score range 1-10; higher scores indicating higher work ability
Pittsburgh Sleep Quality Index (PSQI) | Baseline + 12 weeks
  Sleep Quality (Questionnaire); score range from 0 to 21; lower scores indicating healthier sleep quality
Falls Efficacy Scale (FES) | Baseline + 12 weeks
  Fall Risk Assessment (Questionnaire); score range from 16 to 64; higher values indicate less fall-related self-efficacy (and more concern about falling).

CONTACTS AND LOCATIONS:
Overall Officials: Richard Crevenna, Prof. MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Radocha J, Hajek R, Brozova L, Pour L, Spicka I, Minarik J, Gregora E, Jungova A, Jelinek T, Heindorfer A, Sykora M, Maisnar V. Simplified novel prognostic score for real-life older adults with multiple myeloma-registry-based analysis. Ann Hematol. 2019 Apr;98(4):951-962. doi: 10.1007/s00277-018-3568-2. Epub 2018 Dec 11. PMID 30539278
- [Background] Warren JL, Harlan LC, Stevens J, Little RF, Abel GA. Multiple myeloma treatment transformed: a population-based study of changes in initial management approaches in the United States. J Clin Oncol. 2013 Jun 1;31(16):1984-9. doi: 10.1200/JCO.2012.46.3323. Epub 2013 Apr 8. PMID 23569317
- [Background] Kumar SK, Dispenzieri A, Lacy MQ, Gertz MA, Buadi FK, Pandey S, Kapoor P, Dingli D, Hayman SR, Leung N, Lust J, McCurdy A, Russell SJ, Zeldenrust SR, Kyle RA, Rajkumar SV. Continued improvement in survival in multiple myeloma: changes in early mortality and outcomes in older patients. Leukemia. 2014 May;28(5):1122-8. doi: 10.1038/leu.2013.313. Epub 2013 Oct 25. PMID 24157580
- [Background] Mock V, Pickett M, Ropka ME, Muscari Lin E, Stewart KJ, Rhodes VA, McDaniel R, Grimm PM, Krumm S, McCorkle R. Fatigue and quality of life outcomes of exercise during cancer treatment. Cancer Pract. 2001 May-Jun;9(3):119-27. doi: 10.1046/j.1523-5394.2001.009003119.x. PMID 11879296
- [Background] Crevenna R. Aspects of cancer rehabilitation: an Austrian perspective. Disabil Rehabil. 2020 Jan;42(1):1. doi: 10.1080/09638288.2018.1522554. Epub 2019 Jan 27. No abstract available. PMID 30686037
- [Background] Crevenna R. Cancer rehabilitation and palliative care--two important parts of comprehensive cancer care. Support Care Cancer. 2015 Dec;23(12):3407-8. doi: 10.1007/s00520-015-2977-1. Epub 2015 Oct 6. No abstract available. PMID 26441078
- [Background] Schmitz KH, Courneya KS, Matthews C, Demark-Wahnefried W, Galvao DA, Pinto BM, Irwin ML, Wolin KY, Segal RJ, Lucia A, Schneider CM, von Gruenigen VE, Schwartz AL; American College of Sports Medicine. American College of Sports Medicine roundtable on exercise guidelines for cancer survivors. Med Sci Sports Exerc. 2010 Jul;42(7):1409-26. doi: 10.1249/MSS.0b013e3181e0c112. PMID 20559064
- [Background] Cenik F, Keilani M, Hasenohrl T, Huber D, Stuhlpfarrer B, Pataraia A, Crevenna R. Relevant parameters for recommendations of physical activity in patients suffering from multiple myeloma : A pilot study. Wien Klin Wochenschr. 2020 Mar;132(5-6):124-131. doi: 10.1007/s00508-019-01582-z. Epub 2019 Nov 29. PMID 31784826
- See also: Austrian Cancer Statistics Plasmocytoma/Myeloma — https://www.statistik.at/web_de/statistiken/menschen_und_gesellschaft/gesundheit/krebserkrankungen/plasmozytom_myelom/index.html